CLINICAL TRIAL: NCT05442346
Title: an Open Label Trial of Evaluation of the Safety and Efficacy of Treatment With γ-globin Reactivated Autologous Hematopoietic Stem Cells in Subjects With β-thalassemia Major
Brief Title: Safety and Efficacy Evaluation of γ-globin Reactivated Autologous Hematopoietic Stem Cells
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bioray Laboratories (Industry)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-BRL-103
Record Dates: First submitted 2021-09-23; First posted 2022-07-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-07

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- γ-globin reactivated autologous hematopoietic stem cells (Experimental): each subject will accept one dose of γ-globin reactivated autologous hematopoietic stem cells
  Interventions: Biological: γ-globin reactivated autologous hematopoietic stem cells

INTERVENTIONS:
Biological: γ-globin reactivated autologous hematopoietic stem cells — gene edited autologous hematopoietic stem cells with γ-globin expression; BRL-103

SUMMARY:
This is a single arm, open label, single-dose, phase 1/2 study in up to 5 participants with β-thalassemia major.The study will evaluate the safety and efficacy of the treatment with γ-globin reactivated autologous hematopoietic stem cells in subjects with β-thalassemia major.

DETAILED DESCRIPTION:
γ-globin reactivated autologous hematopoietic stem cells will be manufactured using Glycosylase Base Editors. Subject participation for this study will be 2 year. Subjects who enroll in this study will be asked to participate in a subsequent long-term follow up study that will monitor the safety and efficacy of the treatment they receive for up to 15 years post-transplant.

ELIGIBILITY:
Key inclusion criteria:

* Fully understand and voluntarily sign informed consent. 3-35years old. At least one legal guardian and/or Subjects to sign informed consent.
* Clinically diagnosed as β-thalassemia major, phenotypes including β0β0, β+β+、β

  +β0, βEβ0 genotype.
* Subjects with no affection with EBV, HIV, CMV, TP, HAV, HBV and HCV.
* Subjects body condition eligible for autologous stem cell transplant.

Key exclusion criteria:

* Subjects acceptable for allogeneic hematopoietic stem cell transplantation and have an available fully matched related donor.
* Active bacterial, viral, or fungal infection.
* Treated with erythropoietin prior 3 months.
* Immediate family member with any known hematological tumor.
* Subjects with severe psychiatric disorders to be unable to cooperate.
* Recently diagnosed as malaria.
* History of complex autoimmune disease.
* Persistent aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin value >3 X the upper limit of normal (ULN).
* Subjects with severe heart, lung and kidney diseases.
* With serious iron overload, serum ferritin>5000mg/ml.
* Any other condition that would render the subject ineligible for HSCT, as determined by the attending transplant physician or Investigator.
* Subjects who are receiving treatment from another clinical study, or have received another gene therapy.
* Subjects or guardians had resisted the guidance of the attending doctor.
* Subjects whom the investigators do not consider appropriate for participating in this clinical study

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-09-08 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving successful neutrophil engraftment within 42 days after BRL-103 infusion | From 12 months to 24 months post transplant
Time to neutrophil engraftment | From 12 months to 24 months post transplant
Time to platelet engraftment | From 12 months to 24 months post transplant
Frequency and severity of adverse events through 100 days after BRL-103 Infusion | From 12 months to 24 months post transplant
Proportion of subjects achieving sustained transfusion reduction for at least 3 months (TR3) | From 12 months to 24 months post transplant
  TR3 was defined as at least a 50% reduction in monthly red blood cell transfusion volume and transfusion frequency compared to baseline for at least 3 months

SECONDARY OUTCOMES:
Proportion of subjects achieving sustained transfusion independence for at least 3 months (TI3) | From 12 months to 24 months post transplant
  Routine transfusion without disease related and with Hb ≥ 90 g/L for at least 3 months
Proportion of subjects achieving TR6 | From 12 months to 24 months post transplant
Proportion of subjects achieving TR12 | From 12 months to 24 months post transplant
Proportion of subjects achieving sustained transfusion independence for at least 6 months (TI6) | From 12 months to 24 months post transplant
Proportion of subjects achieving sustained transfusion independence for at least 12 months (TI12) | From 12 months to 24 months post transplant
Incidence of transplant related mortality (TRM) within 100 days and within 1 year | From 12 months to 24 months post transplant
Frequency, severity, and relationship to BRL-103 of adverse events over two years following BRL-103 infusion. | From 12 months to 24 months post transplant
All-cause mortality | From 12 months to 24 months post transplant
Proportion of alleles with intended genetic modification present in peripheral blood leukocytes over time | From 12 months to 24 months post transplant
Fetal hemoglobin concentration (pre-transfusion) over time | From 12 months to 24 months post transplant
Total hemoglobin concentration (pre-transfusion) over time | From 12 months to 24 months post transplant
Change in serum ferritin level from baseline over time | From 12 months to 24 months post transplant

OTHER OUTCOMES:
Changes in the proportion of red blood cells expressing HbF in the blood circulation | From 12 months to 24 months post transplant
LDH levels over time | From 12 months to 24 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: lai yongrong, PhD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- Shanghai Bioray Laboratories Inc, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
clinical study protocol will be shared after Estimated Primary Completion Date
Supporting Information: Study Protocol
Time Frame: data will be available before 2023.10.1, one week long
Access Criteria: university and institute